CLINICAL TRIAL: NCT02851498
Title: Use of Novel High-protein Food Products to Reduce Insulin Resistance in Adults With an Elevated Triglyceride/HDL Ratio
Brief Title: Use of Novel High-protein Food Products To Reduce Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Inflammation Research Foundation (Unknown)
Responsible Party: Principal Investigator, Carol Johnston, Professor, Arizona State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: ArizonaSU2
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Edible Grain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Novel high-protein pasta and cereal (Experimental): High-protein pasta (orzo and fusilli) enriched with gluten and egg white protein (%energy: 27/30/43 for protein/fat/carbohydrate) and high-protein flaked breakfast cereal enriched with gluten (%energy: 30/35/35 for protein/fat/carbohydrate) were manufactured by Zone Inc.(Boston, MA). The study foods provided an average of 945 kcal/day (one aliquot of cereal and two pasta dishes daily). Pasta meals were prepared in a metabolic kitchen and were identical in appearance and basic taste as control meals.
  Interventions: Other: Food product: high-protein pasta and cereal
- Control pasta and cereal (Sham Comparator): Commercial gluten-free pasta (Barcilla orzo and fusilli; %energy: 13/24/63 for protein/fat/carbohydrate) and commercial flaked cereal (Post Honey Bunches of Oats; %energy: 6/18/76 for protein/fat/carbohydrate) were used as the control foods. The study foods provided an average of 945 kcal/day (one aliquot of cereal and two pasta dishes daily). Pasta meals were prepared in a metabolic kitchen and were identical in appearance and basic taste as experimental foods.
  Interventions: Other: Food product: high-protein pasta and cereal

INTERVENTIONS:
Other: Food product: high-protein pasta and cereal

SUMMARY:
This controlled weight loss trial in adults at cardiometabolic risk (elevated triglyceride/HDL ratio) followed a randomized, cross-over design and utilized novel, high-protein pasta and cereal to examine the physiological impact of stealth substitution of dietary carbohydrate with protein derived from soy concentrates, wheat protein isolates, and dried egg whites. Pasta dishes were prepared using high-protein orzo and fusilli pasta (Zone PastaRxTM) or conventional, gluten-free pasta, and high-protein flaked cereal (ZoneTM cereal) was matched with conventional flaked cereal. Participants were instructed to follow an energy restricted diet (-500 kcal/d) and incorporate a test food into each of three meals over a 24-hour period. The diet-induced changes in body mass and lean body mass were tracked as well as changes in in insulin sensitivity and common blood biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* 20-75 years of age
* BMI 23-42 kg/m2

Exclusion Criteria:

* food allergies
* diet restrictions (e.g., vegetarian, gluten or lactose intolerant)
* insulin use
* cigarette use
* active disease states including diagnosed diabetes
* anticipated changes to diet or physical activity levels
* recent weight gain or loss (±10 pounds)
* current or recent pregnancy or lactation
* prescription medication use by participants was allowed if use had been consistent

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Insulin resistance | 6 weeks
  Change in insulin resistance
Body composition | 6 weeks
  Change in body composition

IPD SHARING:
Plan to Share IPD: Undecided